CLINICAL TRIAL: NCT06208306
Title: A Double-blinded Extension Study to Evaluate the Long-term Safety and Tolerability of Itepekimab in Patients With Chronic Obstructive Pulmonary Disease (COPD) Who Participated in Either EFC16750 or EFC16819 Clinical Studies
Brief Title: A Study to Investigate Long-term Safety and Tolerability of Itepekimab in Participants With COPD
Acronym: AERIFY-4
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LTS18133; U1111-1295-3333 (Registry Identifier: ICTRP); 2023-508085-15-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — itepekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Itepekimab Q2W (Experimental): Subcutaneous (SC) administration of Itepekimab every 2 weeks (Q2W) for up to 52 weeks
  Interventions: Drug: Itepekimab (SAR440340)
- Itepekimab Q4W (Experimental): SC administration of Itepekimab every 4 weeks (Q4W) for up to 52 weeks, with alternating SC administration of matching placebo at the 2-week interval between active IMP
  Interventions: Drug: Itepekimab (SAR440340); Drug: Placebo

INTERVENTIONS:
Drug: Itepekimab (SAR440340) — Pharmaceutical form:solution for injection in pre-filled syringe Route of administration:subcutaneous
  Other Names: REGN3500
Drug: Placebo — Pharmaceutical form:solution for injection in pre-filled syringe Route of administration:subcutaneous
  Arms: Itepekimab Q4W

SUMMARY:
This is a parallel, double blind, Phase 3, 2-arm study that is designed to provide additional safety information, assess the durability of treatment response, and provide additional PK and immunogenicity assessments.

The primary purpose of this study is to evaluate safety and tolerability of both itepekimab SC Q2W or itepekimab SC Q4W in participants with COPD having completed the treatment period of the clinical studies EFC16750 or EFC16819. A secondary purpose of this study is to provide efficacy outcomes beyond the treatment period of the parent trials EFC16750 and EFC16819.

Study details include:

* The study duration will be up to 72 weeks
* The treatment duration will be up to 52 weeks
* A follow-up period of 20 weeks will be conducted
* The number of on-site visits will be 7 and the number of phone contacts will be 5

ELIGIBILITY:
Inclusion Criteria:

- Patients with COPD who completed the treatment period in a previous itepekimab COPD Phase 3 clinical study (ie, EFC16750 or EFC16819) and for which an end-of-treatment (EOT) visit occurred no later than 3 days before the enrolment visit of this study.

Exclusion Criteria:

* Diagnosis of a malignancy during parent study, except a squamous or basal cell carcinoma of the skin
* Any opportunistic infection during the parent study, such as tuberculosis (TB) or other infections whose nature or course may suggest an immunocompromised status
* Anaphylactic reactions or systemic allergic reactions that are related to IMP and require treatment during the parent study
* Any situation that led to a permanent premature IMP discontinuation in parent trials

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AEs, AESIs, SAEs, and AEs leading to permanent treatment discontinuation | Baseline up to Week 72
  All AEs (serious or nonserious) will be collected from the signing of the informed consent form (ICF) until the end of study visit

SECONDARY OUTCOMES:
Functional itepekimab concentrations in serum | Baseline up to Week 52
Incidence of treatment-emergent (TE) anti-drug antibody responses | Baseline up to Week 72
Annualized rate of moderate-to-severe acute exacerbation of COPD (AECOPD) | Baseline up to Week 52
Annualized rate of severe AECOPD | Baseline up to Week 52
Time to first moderate-to-severe AECOPD | Baseline up to Week 52
Time to first severe AECOPD | Baseline up to Week 52
Change from baseline of the parent studies (EFC16750, EFC16819): Pre-BD and post-BD FEV1 | Baseline of the parent studies (EFC16750,EFC16819) up to Week 52
  FEV1 is force expiratory volume in 1 second
Change from baseline of the parent studies (EFC16750, EFC16819): SGRQ total score and domain scores | Baseline of the parent studies (EFC16750,EFC16819) up to Week 52
  The St. George's Respiratory Questionnaire (SGRQ) is a 50-item questionnaire designed to measure and quantify health status in adult participants with chronic airflow limitation.
Change from baseline of the parent studies (EFC16750, EFC16819): EQ-5D-5L single index score | Baseline of the parent studies (EFC16750,EFC16819) up to Week 52
  The European Quality of Life 5 Dimensions 5 Level Version (EQ 5D 5L) is a standardized health-related quality-of-life (HRQoL) questionnaire which consists of a descriptive system and the EuroQol visual analog scale (EQ-VAS).
Change from baseline of the parent studies (EFC16750, EFC16819): EQ-VAS | Baseline of the parent studies (EFC16750,EFC16819) up to Week 52
  The EuroQol visual analog scale (EQ VAS) records the participant's self-rated health on a vertical VAS.
Change from Week 0 for CASA-Q | Baseline up to Week 52
  The cough and sputum assessment questionnaire (CASA-Q) was developed for use in COPD and chronic (non-obstructive) bronchitis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (223):
- United States (64):
  - Chandler Clinical Research Trials- Site Number : 8401034, Chandler, Arizona
  - Noble Clinical Research Site Number : 8401182, Tucson, Arizona
  - Tucson Clinical Research Institute- Site Number : 8401431, Tucson, Arizona
  - IMAX Clinical Trials- Site Number : 8401419, La Palma, California
  - Antelope Valley Clinical Trials Site Number : 8401003, Lancaster, California
  - Downtown L.A. Research Center- Site Number : 8401027, Los Angeles, California
  - Allianz Research Institute CO Site Number : 8402061, Aurora, Colorado
  - Alpine Clinical Research Center - Boulder - 47th Street- Site Number : 8401180, Boulder, Colorado
  - Helix Biomedics- Site Number : 8402049, Boynton Beach, Florida
  - Beautiful Minds Clinical Research Center Site Number : 8401201, Cutler Bay, Florida
  - Omega Research Consultants - Debary - North Charles Richard Beall Boulevard- Site Number : 8402031, DeBary, Florida
  - Science Connections, LLC Site Number : 8402045, Doral, Florida
  - Direct Helpers Research Center- Site Number : 8402065, Hialeah, Florida
  - Premier Medical Associates Site Number : 8401388, Lady Lake, Florida
  - Advanced Pulmonary Research Institute Site Number : 8402018, Loxahatchee Groves, Florida
  - Finlay Medical Research- Site Number : 8402007, Miami, Florida
  - Elite Clinical Research - Miami- Site Number : 8402009, Miami, Florida
  - DL Research Solutions- Site Number : 8401033, Miami, Florida
  - My Community Research Center Site Number : 8402060, Miami, Florida
  - Phoenix Medical Research - Miami - 24th Street- Site Number : 8402019, Miami, Florida
  - Research Institute of South Florida- Site Number : 8401006, Miami, Florida
  - Reed Medical Research Site Number : 8401032, Miami, Florida
  - High Quality Research Site Number : 8401406, Miami, Florida
  - Deluxe Health Center Site Number : 8401188, Miami Lakes, Florida
  - Renstar Medical Research - Ocala - Northeast 1st Avenue- Site Number : 8402015, Ocala, Florida
  - Heuer M.D. Research- Site Number : 8402016, Orlando, Florida
  - Florida Institute for Clinical Research Site Number : 8401013, Orlando, Florida
  - Oviedo Medical Research Site Number : 8402026, Oviedo, Florida
  - Innovation Medical Research Center - Palmetto Bay- Site Number : 8402067, Palmetto Bay, Florida
  - Pines Care Research Center- Site Number : 8402056, Pembroke Pines, Florida
  - Tellabio International Research Services Site Number : 8401411, Pembroke Pines, Florida
  - Clinical Research of West Florida - Tampa - North Howard Avenue- Site Number : 8402008, Tampa, Florida
  - Appalachian Clinical Research Site Number : 8400024, Calhoun, Georgia
  - Private Practice - Dr. David Kavtaradze- Site Number : 8401029, Cordele, Georgia
  - Alpha Clinical Research Group - Dunwoody- Site Number : 8401190, Dunwoody, Georgia
  - Covenant Pulmonary Critical Care Site Number : 8401183, East Point, Georgia
  - OSF Saint Fracis Medical Center- Site Number : 8402024, Peoria, Illinois
  - Benchmark Research - Covington- Site Number : 8401193, Covington, Louisiana
  - Care Access - Shreveport- Site Number : 8402047, Shreveport, Louisiana
  - Private Practice - Dr. Paul Shapero- Site Number : 8401016, Bangor, Maine
  - Care Access - Boston- Site Number : 8402276, Boston, Massachusetts
  - Revive Research Institute - Lathrup Village- Site Number : 8402186, Lathrup Village, Michigan
  - Pulmonary and Medicine Associates- Site Number : 8401403, Warren, Michigan
  - Hannibal Regional Healthcare System-HRMG-Hannibal Site Number : 8401383, Hannibal, Missouri
  - Midwest Chest Consultants- Site Number : 8401002, Saint Charles, Missouri
  - Washington University- Site Number : 8402035, St Louis, Missouri
  - Henderson Clinical Trials Site Number : 8401365, Henderson, Nevada
  - VA Western New York Healthcare System Site Number : 8402050, Buffalo, New York
  - Schenectady Pulmonary and Critical Care Associates - Schenectady Main Office- Site Number : 8402029, Schenectady, New York
  - East Carolina University- Site Number : 8401022, Greenville, North Carolina
  - Advanced Respiratory and Sleep Medicine - Huntersville- Site Number : 8400022, Huntersville, North Carolina
  - OK Clinical Research- Site Number : 8402001, Edmond, Oklahoma
  - Clinical Research Associates of Central PA - Dubois- Site Number : 8401023, DuBois, Pennsylvania
  - Allegheny General Hospital- Site Number : 8402058, Pittsburgh, Pennsylvania
  - MedTrial- Site Number : 8402048, Columbia, South Carolina
  - Clinical Research of Rock Hill Site Number : 8401008, Rock Hill, South Carolina
  - REX Clinical Trials - Beaumont- Site Number : 8401371, Beaumont, Texas
  - South Texas Medical Research Institute - TTS Research- Site Number : 8402012, Boerne, Texas
  - ClinRx Research - Carrollton- Site Number : 8401021, Carrollton, Texas
  - Corsicana Medical Research- Site Number : 8401018, Corsicana, Texas
  - The Methodist Hospital Research Institute Site Number : 8401194, Houston, Texas
  - Metroplex Pulmonary and Sleep Center Site Number : 8401015, McKinney, Texas
  - Clear Lake Specialties Research Center, PLLC Site Number : 8401025, Webster, Texas
  - Rheumatology & Pulmonary Clinic- Site Number : 8402053, Beckley, West Virginia
- Argentina (12):
  - Investigational Site Number : 0320012, Berazategui, Buenos Aires
  - Investigational Site Number : 0320013, La Plata, Buenos Aires
  - Investigational Site Number : 0320003, Rosario, Santa Fe Province
  - Investigational Site Number : 0320007, Rosario, Santa Fe Province
  - Investigational Site Number : 0320008, Rosario, Santa Fe Province
  - Investigational Site Number : 0320011, Rosario, Santa Fe Province
  - Investigational Site Number : 0320010, Buenos Aires
  - Investigational Site Number : 0320005, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320006, Buenos Aires
  - Investigational Site Number : 0320009, Buenos Aires
  - Investigational Site Number : 0320004, Mendoza
- Brazil (13):
  - Centro de Diagnostico e Pesquisa da Osteoporose do Espirito Santo- Site Number : 0760009, Vitória, Espírito Santo
  - Serviços Especializados em Reumatologia- Site Number : 0760020, Salvador, Estado de Bahia
  - Centro De Cardiologia Clinica E Pesquisa- Site Number : 0760018, Brasília, Federal District
  - Santa Casa de Misericordia de Belo Horizonte- Site Number : 0760014, Belo Horizonte, Minas Gerais
  - Centro de Estudos em Terapias Inovadoras- Site Number : 0760012, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre- Site Number : 0760001, Porto Alegre, Rio Grande do Sul
  - Instituto Ceos Site Number : 0760021, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS - Porto Alegre - Avenida Ipiranga- Site Number : 0760007, Porto Alegre, Rio Grande do Sul
  - WM Pesquisas Clínicas em Doenças Respiratórias- Site Number : 0760006, Porto Alegre, Rio Grande do Sul
  - Universidade Estadual Paulista - Faculdade de Medicina de Botucatu- Site Number : 0760005, Botucatu, São Paulo
  - Hospital e Maternidade Celso Pierro - PUC-Campinas- Site Number : 0760010, Campinas, São Paulo
  - Centro Multidisciplinar de Estudos Clínicos- Site Number : 0760015, São Bernardo do Campo, São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo- Site Number : 0760013, São Paulo
- Bulgaria (11):
  - Investigational Site Number : 1000004, Gabrovo
  - Investigational Site Number : 1000007, Haskovo
  - Investigational Site Number : 1000018, Rousse
  - Investigational Site Number : 1000010, Rousse
  - Investigational Site Number : 1000016, Sofia
  - Investigational Site Number : 1000001, Sofia
  - Investigational Site Number : 1000009, Sofia
  - Investigational Site Number : 1000017, Stara Zagora
  - Investigational Site Number : 1000003, Stara Zagora
  - Investigational Site Number : 1000013, Veliko Tarnovo
  - Investigational Site Number : 1000006, Vidin
- Canada (8):
  - Investigational Site Number : 1240006, Sherwood Park, Alberta
  - Investigational Site Number : 1240021, Ajax, Ontario
  - Investigational Site Number : 1240009, Toronto, Ontario
  - Investigational Site Number : 1240022, Windsor, Ontario
  - Investigational Site Number : 1240018, Windsor, Ontario
  - Investigational Site Number : 1240004, Sherbrooke, Quebec
  - Investigational Site Number : 1240001, Trois-Rivières, Quebec
  - Investigational Site Number : 1240002, Victoriaville, Quebec
- Chile (7):
  - Investigational Site Number : 1520008, Valdivia, Los Ríos Region
  - Investigational Site Number : 1520006, Talca, Maule Region
  - Investigational Site Number : 1520007, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Quillota, Región de Valparaíso
- China (16):
  - Investigational Site Number : 1560012, Beijing
  - Investigational Site Number : 1560004, Changchun
  - Investigational Site Number : 1560001, Chengdu
  - Investigational Site Number : 1560018, Haikou
  - Investigational Site Number : 1560016, Hefei
  - Investigational Site Number : 1560017, Hohhot
  - Investigational Site Number : 1560002, Jinan
  - Investigational Site Number : 1560014, Nanchang
  - Investigational Site Number : 1560019, Pingxiang
  - Investigational Site Number : 1560020, Shanghai
  - Investigational Site Number : 1560006, Shanghai
  - Investigational Site Number : 1560008, Shenyang
  - Investigational Site Number : 1560005, Wuhan
  - Investigational Site Number : 1560011, Xiangtan
  - Investigational Site Number : 1560007, Xuzhou
  - Investigational Site Number : 1560015, Yangzhou
- Czechia (2):
  - Investigational Site Number : 2030003, Havlíčkův Brod
  - Investigational Site Number : 2030001, Jindřichův Hradec
- Investigational Site Number : 2330001, Tartu, Estonia
- France (2):
  - Investigational Site Number : 2500001, Lyon
  - Investigational Site Number : 2500004, Reims
- Georgia (4):
  - Investigational Site Number : 2680006, Batumi
  - Investigational Site Number : 2680002, Tbilisi
  - Investigational Site Number : 2680003, Tbilisi
  - Investigational Site Number : 2680001, Tbilisi
- Germany (8):
  - Investigational Site Number : 2760006, Bendorf
  - Investigational Site Number : 2760010, Berlin
  - Investigational Site Number : 2760005, Frankfurt
  - Investigational Site Number : 2760008, Leipzig
  - Investigational Site Number : 2760007, Leipzig
  - Investigational Site Number : 2760003, Lübeck
  - Investigational Site Number : 2760001, Mainz
  - Investigational Site Number : 2760011, Rosenheim
- Greece (2):
  - Investigational Site Number : 3000008, Palaió Fáliro
  - Investigational Site Number : 3000002, Thessaloniki
- Hungary (5):
  - Investigational Site Number : 3480009, Budapest
  - Investigational Site Number : 3480001, Gödöllő
  - Investigational Site Number : 3480004, Hajdúnánás
  - Investigational Site Number : 3480002, Mosonmagyaróvár
  - Investigational Site Number : 3480003, Püspökladány
- India (11):
  - Investigational Site Number : 3560001, Calicut
  - Investigational Site Number : 3560006, Chandigarh
  - Investigational Site Number : 3560005, Hyderabad
  - Investigational Site Number : 3560009, Jaipur
  - Investigational Site Number : 3560004, Jaipur
  - Investigational Site Number : 3560012, Kanpur
  - Investigational Site Number : 3560010, Nagpur
  - Investigational Site Number : 3560011, Nagpur
  - Investigational Site Number : 3560007, Nagpur
  - Investigational Site Number : 3560003, Nagpur
  - Investigational Site Number : 3560013, Pune
- Israel (8):
  - Investigational Site Number : 3760008, Haifa
  - Investigational Site Number : 3760003, Jerusalem
  - Investigational Site Number : 3760002, Jerusalem
  - Investigational Site Number : 3760006, Kefar Sava
  - Investigational Site Number : 3760001, Petah Tikva
  - Investigational Site Number : 3760009, Ramat Gan
  - Investigational Site Number : 3760004, Rehovot
  - Investigational Site Number : 3760007, Tel Aviv
- Investigational Site Number : 3800001, Ferrara, Italy
- Japan (9):
  - Investigational Site Number : 3920008, Nagoya, Aichi-ken
  - Investigational Site Number : 3920002, Kurume, Fukuoka
  - Investigational Site Number : 3920007, Kure, Hiroshima
  - Investigational Site Number : 3920006, Himeji, Hyōgo
  - Investigational Site Number : 3920009, Yokohama, Kanagawa
  - Investigational Site Number : 3920001, Matsusaka, Mie-ken
  - Investigational Site Number : 3920005, Kiyose, Tokyo
  - Investigational Site Number : 3920003, Fukuoka
  - Investigational Site Number : 3920004, Tokyo
- Investigational Site Number : 4400002, Kaunas, Lithuania
- Investigational Site Number : 4840007, Durango, Mexico
- Investigational Site Number : 5280001, Breda, Netherlands
- Investigational Site Number : 5780001, Lørenskog, Norway
- Poland (2):
  - Investigational Site Number : 6160001, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6160002, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- Investigational Site Number : 6200006, Porto, Portugal
- Investigational Site Number : 6420002, Cluj-Napoca, Romania
- Slovakia (3):
  - Investigational Site Number : 7030002, Humenné
  - Investigational Site Number : 7030004, Prešov
  - Investigational Site Number : 7030003, Spišská Nová Ves
- South Africa (4):
  - Investigational Site Number : 7100004, Benoni
  - Investigational Site Number : 7100001, Durban
  - Investigational Site Number : 7100006, Durban
  - Investigational Site Number : 7100005, Durban
- South Korea (2):
  - Investigational Site Number : 4100002, Wŏnju, Gangwon-do
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
- Spain (8):
  - Investigational Site Number : 7240014, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240006, Sant Boi de Llobregat, Catalunya [Cataluña]
  - Investigational Site Number : 7240008, Pozuelo de Alarcón, Madrid
  - Investigational Site Number : 7240003, Madrid
  - Investigational Site Number : 7240007, Madrid
  - Investigational Site Number : 7240001, Málaga
  - Investigational Site Number : 7240004, Palma
  - Investigational Site Number : 7240012, Zaragoza
- Taiwan (3):
  - Investigational Site Number : 1580005, Kaohsiung City
  - Investigational Site Number : 1580006, Taichung
  - Investigational Site Number : 1580003, Taipei
- Turkey (Türkiye) (4):
  - Investigational Site Number : 7920002, Akdeniz
  - Investigational Site Number : 7920007, Ankara
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920006, Kırıkkale
- United Kingdom (7):
  - Investigational Site Number : 8260004, Portsmouth, Hampshire
  - Investigational Site Number : 8260002, Chertsey, Surrey
  - Investigational Site Number : 8260003, Bradford
  - Investigational Site Number : 8260014, Hounslow
  - Investigational Site Number : 8260005, Liverpool
  - Investigational Site Number : 8260010, London
  - Investigational Site Number : 8260008, Milton Keynes

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org